CLINICAL TRIAL: NCT00437892
Title: The Effect of Statins on D-dimer Levels in Patients With a Previous Venous Thromboembolic Event
Brief Title: Statins to Reduce D-dimer Levels in Patients With Venous Thrombosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Competitive trials and slow recruitment rate
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Walter Ageno, Associate Professor of Internal Medicine, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7948
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Venous Thromboembolism; Hypercholesterolemia
Keywords: Statins; secondary prevention; venous thromboembolism; d-dimer
MeSH Terms: conditions — Venous Thromboembolism; Hypercholesterolemia | interventions — Atorvastatin; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin and lipid lowering diet (Experimental)
  Interventions: Drug: atorvastatin; Behavioral: diet
- lipid lowering diet (Active Comparator)
  Interventions: Behavioral: diet

INTERVENTIONS:
Drug: atorvastatin — tablets, 40 mg day, 3 months
  Arms: Atorvastatin and lipid lowering diet
Drug: atorvastatin — tablets, 40 mg once daily
  Arms: Atorvastatin and lipid lowering diet
Behavioral: diet — daily
  Arms: lipid lowering diet
Behavioral: diet — daily diet

SUMMARY:
Elevated levels of D-dimer, a marker of procoagulant state, have been identified as a marker of an increased risk of recurrent VTE. Statins have proven antithrombotic properties, as suggested by the reduction of several prothrombotic markers, including D-dimer, in patients at high risk of arterial thrombosis. Such antithrombotic properties could also be observed in patients at high risk of venous thrombosis. Aim of the study is to assess the effect of statins on D-dimer levels in patients with previous VTE after oral anticoagulant treatment withdrawal.

DETAILED DESCRIPTION:
Patients with a single episode of idiopathic VTE (either DVT or pulmonary embolism) who received at least 6 months of adequate treatment with oral anticoagulants, for whom treatment withdrawal is planned, and with LDL cholesterol levels of equal to or greater than 130 mg/dL will be randomized to either atorvastatin, 40 mg, 1 tablet daily and lipid lowering diet or lipid lowering diet for 3 months. On the day of oral anticoagulant treatment withdrawal (Day 0), enrolled patients will undergo measurement of plasma D-dimer. At 30 days ± 3 (Day 30), patients will undergo measurement of D-dimer, CK, LDH, ALAT e ASAT and clinical evaluation. At 90 days ± 7 (Day 90), patients will undergo measurement of D-dimer, total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides ed clinical evaluation, CK, LDH, ALAT e ASAT. At 6 months ± 1 (Day 180), patients will undergo clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a single episode of idiopathic VTE (either DVT or pulmonary embolism) who received at least 6 months of adequate treatment with oral anticoagulants, for whom treatment withdrawal is planned, and with LDL cholesterol levels of equal to or greater than 130 mg/dL.

Exclusion Criteria:

* Age below 18 years,
* Pregnancy or puerperium,
* Active malignancy,
* Need for other anticoagulant treatments (unfractionated heparin, low molecular weight heparin),
* Presence of transient risk factors for VTE [recent (< 3 months) surgery,
* Trauma,
* Fractures,
* Acute medical disease with immobilization,
* Pregnancy or use of oral contraceptives],
* Contraindications to statin therapy,
* Chronic renal failure (defined by creatinine clearance < 30 mL/min),
* Ongoing treatment with statins or fibrates,
* Major indication to statin therapy [history of cardiovascular disease, diabetes, elevated cardiovascular risk according to the ATP III criteria(19)],
* Life expectancy of less than 6 months,
* Geographic inaccessibility,
* Concomitant enrolment in another clinical trial,
* Refused informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
proportion of patients with elevated D-dimer at day 90 | 3 months

SECONDARY OUTCOMES:
proportion of patients with elevated D-dimer levels at Day 30; | 1 month
proportion of patients with elevated D-dimer levels at Day 0 and subsequent normalization of D-dimer levels at Day 30 and Day 90; | 3 months
proportion of patients with recurrent VTE | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ageno, Principal Investigator — Università degli Studi dell'Insubria; Gualtiero Palareti, Principal Investigator — University of Bologna; Davide Imberti, Principal Investigator — Piacenza Hospital
Locations (3):
- Italy (3):
  - University of Bologna, Bologna
  - Ospedale di Piacenza, Piacenza
  - University Of Insubria, Varese

REFERENCES:
- [Background] Palareti G, Cosmi B, Legnani C, Tosetto A, Brusi C, Iorio A, Pengo V, Ghirarduzzi A, Pattacini C, Testa S, Lensing AW, Tripodi A; PROLONG Investigators. D-dimer testing to determine the duration of anticoagulation therapy. N Engl J Med. 2006 Oct 26;355(17):1780-9. doi: 10.1056/NEJMoa054444. PMID 17065639
- [Background] Squizzato A, Romualdi E, Ageno W. Why should statins prevent venous thromboembolism? A systematic literature search and a call for action. J Thromb Haemost. 2006 Sep;4(9):1925-7. doi: 10.1111/j.1538-7836.2006.02030.x. No abstract available. PMID 16961599